CLINICAL TRIAL: NCT04368559
Title: A Phase 3, Multicenter, Randomized, Double-Blind Study of the Efficacy and Safety of Rezafungin for Injection Versus the Standard Antimicrobial Regimen to Prevent Invasive Fungal Diseases in Adults Undergoing Allogeneic Blood and Marrow Transplantation (The ReSPECT Study)
Brief Title: Study of Rezafungin Compared to Standard Antimicrobial Regimen for Prevention of Invasive Fungal Diseases in Adults Undergoing Allogeneic Blood and Marrow Transplantation
Acronym: ReSPECT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CD101.IV.3.08; 2017-004981-85 (EudraCT Number)
Record Dates: First submitted 2020-04-22; First posted 2020-04-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Candidemia; Mycoses; Fungal Infection; Fungemia; Invasive Candidiasis; Pneumocystis; Mold Infection; Invasive Fungal Disease; Prophylaxis of Invasive Fungal Infections; Aspergillus
Keywords: Mycoses; Prophylaxis of Invasive Fungal Infections; Aspergillus; Candidiasis; Candidemia; Candidiasis, Invasive; Fungemia; Sepsis; Blood and Marrow Transplant (BMT); Infection; Invasive Fungal Infections; Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes; Fluconazole; Posaconazole; Caspofungin; Trimethoprim-sulfamethoxazole (TMP/SMX); Echinocandins; Antifungal Agents; 14-alpha Demethylase Inhibitors; Cytochrome P-450 Enzyme Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Steroid Synthesis Inhibitors; Physiological Effects of Drugs; Cytochrome P-450 CYP2C9 Inhibitors; Cytochrome P-450 CYP2C19 Inhibitors; Pneumocystis; Mold Infection; Rezafungin; Anti-Infective Agents
MeSH Terms: conditions — Candidemia; Mycoses; Fungemia; Candidiasis, Invasive; Pneumonia, Pneumocystis; Invasive Fungal Infections; Candidiasis; Sepsis; Infections; Systemic Inflammatory Response Syndrome; Inflammation; Pathologic Processes | interventions — Rezafungin; Injections; posaconazole; Fluconazole; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: Rezafungin for Injection (Experimental): Subjects in Rezafungin treatment group will receive a 400 mg loading dose in Week 1, followed by 200 mg once weekly, for a total of 13 weeks. Subjects will receive oral placebo for standard antimicrobial regimen (SAR) azole prophylaxis and oral placebo for SAR anti-Pneumocystis pneumonia (PCP) prophylaxis in accordance with the respective SAR dosing regimens for each. For subjects who are switched to a SAR IV regimen, oral placebo for SAR azole prophylaxis will be changed to IV placebo. There is no IV option for SAR anti-PCP prophylaxis.
  Interventions: Drug: Rezafungin for Injection; Drug: Intravenous Placebo; Drug: Oral Placebo
- Group 2: Oral Antifungal (Active Comparator): Subjects randomized to the SAR will receive either fluconazole or posaconazole as the first-line SAR as per site's standard practice. Fluconazole will be administered orally at once daily doses of 400 mg for 13 weeks. Posaconazole will be administered orally as 300 mg twice daily on the first day and 300 mg once daily thereafter for 13 weeks. Azole-based antifungal therapy (fluconazole or posaconazole) can be switched from oral therapy to IV therapy if there is oral intolerance, at the discretion of the Investigator.
  Subjects who started on fluconazole SAR may be switched to posaconazole at the discretion of the Investigator if they develop acute clinically significant GVHD; In addition, subjects in the SAR group will receive anti PCP prophylaxis with oral TMP/SMX (80 mg TMP/ 400 mg SMX) once daily. There is no IV option for SAR anti-PCP prophylaxis.
  Interventions: Drug: Posaconazole; Drug: Fluconazole; Drug: Trimethoprim-sulfamethoxazole (TMP/SMX)

INTERVENTIONS:
Drug: Rezafungin for Injection — Intravenous antifungal therapy
  Other Names: Intravenous antifungal therapy
  Arms: Group 1: Rezafungin for Injection
Drug: Posaconazole — Oral antifungal therapy
  Other Names: Noxafil
  Arms: Group 2: Oral Antifungal
Drug: Fluconazole — Oral antifungal therapy
  Other Names: Generic Fluconazole
  Arms: Group 2: Oral Antifungal
Drug: Trimethoprim-sulfamethoxazole (TMP/SMX) — Oral antibacterial therapy
  Other Names: Bactrim; Septra
  Arms: Group 2: Oral Antifungal
Drug: Intravenous Placebo — Normal saline
  Other Names: Placebo Infusion
  Arms: Group 1: Rezafungin for Injection
Drug: Oral Placebo — Microcrystalline cellulose
  Other Names: encapsulated cellulose
  Arms: Group 1: Rezafungin for Injection

SUMMARY:
The purpose of this pivotal study is to determine if intravenous Rezafungin is efficacious and safe in the prevention of invasive fungal diseases when compared to the standard antimicrobial regimen.

DETAILED DESCRIPTION:
A Phase 3, multicenter, prospective, randomized, double-blind, efficacy and safety study of Rezafungin for injection versus the standard antimicrobial regimen for the prevention of invasive fungal diseases in subjects undergoing allogeneic blood and marrow transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Males or females ≥18 years of age.
3. Receiving a human leukocyte antigen (HLA) matched allogeneic peripheral BMT from a family or unrelated donor, HLA-mismatched related or unrelated donor, or haploidentical donor.
4. Diagnosed with 1 of the following underlying diseases:

   1. Acute myeloid leukemia (AML), with or without a history of myelodysplastic syndrome, in first or second complete remission.
   2. Acute lymphoblastic leukemia, in first or second complete remission.
   3. Acute undifferentiated leukemia in first or second remission.
   4. Acute biphenotypic leukemia in first or second complete remission.
   5. Chronic myelogenous leukemia in either chronic or accelerated phase.
   6. One of the following myelodysplastic syndrome(s) defined by the following:

   i. Refractory anemia.

   ii. Refractory anemia with ringed sideroblasts.

   iii. Refractory cytopenia with multilineage dysplasia.

   iv. Refractory cytopenia with multilineage dysplasia and ringed sideroblasts.

   v. Refractory anemia with excess blasts - 1 (5-10% blasts).

   vi. Refractory anemia with excess blasts - 2 (10-20% blasts).

   vii. Myelodysplastic syndrome, unclassified.

   viii. Myelodysplastic syndrome associated with isolated del (5q).

   g. Lymphoma (including Hodgkin's) with chemosensitive disease (i.e., response to chemotherapy) and receiving a related or unrelated donor transplant.

   h. Aplastic anemia.

   i. Primary or secondary myelofibrosis.

   j. Chronic myelomonocytic leukemia.

   k. Chronic lymphocytic leukemia.

   l. Drepanocytosis (sickle cell anemia).

   m. Red blood cell aplasia.

   n. Myeloproliferative disorder, unclassified.

   o. Multiple myeloma (plasma cell myeloma).
5. Receiving myeloablative or reduced-intensity conditioning regimens.
6. Adequate renal and hepatic function prior to initiation of conditioning regimen, therefore between 40 days prior and 10 days prior to BMT, documented as follows:

   1. Hepatic: alanine aminotransferase less than or equal to (≤) 2.5 × upper limit of normal (ULN) and total serum bilirubin ≤1.5 × ULN (excluding Gilbert's Syndrome).
   2. Renal: serum creatinine ≤2 milligrams (mg)/deciliter (dL) and with creatinine clearance (CrCl) greater than or equal to (≥) 30 milliliters (mL)/minute (min) without a history of renal transplant, or undergoing weekly dialysis within 4 weeks of the BMT.
7. Baseline blood samples drawn for Platelia galactomannan enzyme immunoassay (GM EIA) and β-D glucan levels within 15 days before randomization, with results available prior to randomization.
8. Baseline Toxoplasma serologies available within 6 weeks prior to randomization. Subjects with a positive toxoplasma IgG serology at any time prior to randomization do not need to repeat the toxoplasma serologies (IgG and IgM) and will be considered to have a prior history of toxoplasmosis.
9. Baseline glucose-6-phosphate dehydrogenase (G6PD) deficiency determination by the investigator prior to randomization with no known evidence of G6PD deficiency performed any time prior to randomization. If the Investigator assesses the subject as G6PD sufficient, the G6PD test result does not need to be entered into the EDC system.
10. Female subjects of child-bearing potential <2 years post-menopausal (unless surgically sterile) must agree to and comply with using 1 barrier method (e.g., female condom with spermicide) plus one other highly effective method of birth control (e.g., oral contraceptive, implant, injectable, indwelling intrauterine device, vasectomized partner), or sexual abstinence (only possible if it corresponds to the subject's usual lifestyle) while participating in this study, and for 30 days after the last dose of study drug. Male subjects must be vasectomized, abstain from sexual intercourse, or agree to use barrier contraception (condom with spermicide), and agree not to donate sperm while participating in the study and for 120 days from the last IV dose of study drug.

Exclusion Criteria:

1. Diagnosis of AML not in morphological remission.
2. Diagnosis of chemotherapy-resistant lymphoma: a first relapse can occur provided that a second complete remission has occurred.
3. Suspected or diagnosed invasive fungal disease (IFD) within 4 weeks of randomisation.
4. Diagnosed symptomatic heart failure with left ventricular ejection fraction (LVEF) at rest ≤50%, or shortening fraction ≤26%.
5. Personal or family history of Long QT interval on electrocardiogram (ECG) (QT) syndrome or a prolonged QT interval corrected for heart rate by Fridericia's formula (QTcF) (>470 milliseconds [msec] in males and >480 msec in females); or concurrent administration of terfenadine, cisapride, astemizole, erythromycin, pimozide, quinidine, or halofantrine.
6. Diagnosed reduced lung function with either diffusion capacity (corrected for hemoglobin) or forced expiratory volume in 1 second (FEV1) ≤65% of predicted value, or O2 saturation ≤82% on room air.
7. Suspected or documented PCP within 2 years of screening.
8. Positive baseline serum Platelia GM EIA (≥ 0.5) and/or β-D glucan assay (Fungitell ≥80 picograms [pg]/mL or Fujifilm Wako >11 pg/mL) within 15 days prior to the transplant.
9. Receipt of previous allogeneic BMT.
10. Planned receipt of cord blood for transplantation.
11. Planned peripheral blood or marrow autograft.
12. Not applicable to protocol Amendment 6.
13. Grade 2 or higher ataxia, tremor, motor neuropathy, or sensory neuropathy, per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
14. History of severe (Grade ≥3) ataxia, neuropathy or tremors; or a diagnosis of multiple sclerosis or a movement disorder (including Parkinson's disease or Huntington's disease).
15. . .

    1. Planned or ongoing intake at screening of a known severe neurotoxic medication or with a known moderate neurotoxic medication in a patient with ataxia, tremor, motor neuropathy, or sensory neuropathy of CTCAE version 5.0 Grade 1 or higher.
    2. Any contraindication or a medication or supplement known to severely interact with the standard antimicrobial regimen (SAR) as detailed in the US Prescribing Information (USPI) or Summary of Product Characteristics (SmPC) of fluconazole, posaconazole, or TMP/SMX.
16. Known hypersensitivity to Rezafungin for Injection, any echinocandin, fluconazole, posaconazole, other azole antifungal, or to any of their excipients.
17. Known hypersensitivity or inability to receive TMP/SMX or any of its excipients, including but not limited to anaphylaxis, exfoliative skin disorders, or acute porphyria.
18. Recent use of an investigational medicinal product within 28 days or 5 half-lives of the investigational medicinal product, whichever is greater, to prevent overlapping toxicities when this study's investigational product is dosed, or presence of an investigational device at the time of screening. In some cases, use of investigational products may be acceptable in consultation with the Sponsor's Medical Monitor.
19. Known infection with HIV. Subjects with unknown HIV status should be tested for HIV antibodies per standard of care.
20. Pregnant or lactating females.
21. The Principal Investigator (PI) determines that the subject should not participate in the study.
22. Considered unlikely to follow up for 90 days after receipt of the BMT due to logistic concerns (i.e., location relative to transplant center).
23. Known liver cirrhosis, diagnosed according to country or Medical Society specific guidelines and documented in the medical records prior to initiating conditioning regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Noninferior Fungal-Free Survival (US FDA) | Day 90 (±7 days)
  The number of subjects in each treatment group who are fungal-free and survive.
Noninferior Fungal-Free Survival (US FDA) | Day 90 (±7 days)
  The percentage of subjects in each treatment group who are fungal-free and survive.
Superior Fungal-Free Survival (EMA) | Day 90 (±7 days)
  The number of subjects in each treatment group who are fungal-free and survive.
Superior Fungal-Free Survival (EMA) | Day 90 (±7 days)
  The percentage of subjects in each treatment group who are fungal-free and survive.

SECONDARY OUTCOMES:
Compare Discontinuation for Toxicity or Intolerance | Day 90 (±7 days)
  The number of subjects that discontinued Rezafungin for Injection compared to the standard antimicrobial regimen (SAR) secondary to toxicity or intolerance.
Compare Discontinuation for Toxicity or Intolerance | Day 90 (±7 days)
  The percentage of subjects that discontinued Rezafungin for Injection compared to the standard antimicrobial regimen (SAR) secondary to toxicity or intolerance.
Compare Proven and Probable IFD | Day 90 (±7 days)
  The number of subjects in each treatment group who have proven and probable IFD including the number of invasive infections from Candida spp., Aspergillus spp., and Pneumocystis jirovecii.
Compare Proven and Probable IFD | Day 90 (±7 days)
  The percentage of subjects in each treatment group who have proven and probable IFD including the number of invasive infections from Candida spp., Aspergillus spp., and Pneumocystis jirovecii.
Compare Fungal-Free Survival with or without a Diagnosis of Clinically Significant GVHD | Day 90 (±7 days)
  The number of subjects in each treatment group who are fungal-free survival with or without a diagnosis of clinically significant GVHD.
Compare Fungal-Free Survival with or without a Diagnosis of Clinically Significant GVHD | Day 90 (±7 days)
  The percentage of subjects in each treatment group who are fungal-free survival with or without a diagnosis of clinically significant GVHD.
Compare Time to IFD, or Death | Day 90 (±7 days)
  Evaluate time to IFD (proven or probable IFD) or death in subjects randomized to Rezafungin for Injection compared to the standard antimicrobial regimen (SAR).
Compare Mortality | Day 1 through follow-up visit (Day 120)
  Evaluate overall mortality and attributable mortality, with and without adjustment for patient comorbidity indices, in subjects randomized to Rezafungin for Injection compared to the SAR.
Incidence of Treatment Emergent Adverse Events [Safety and Tolerability] | Day 1 through follow-up visit (Day 120)
  The number of subjects with incidence of treatment emergent adverse events based on clinical chemistry, hematology and urine analysis laboratory test, vital sign, physical exams and ECG abnormalities.

OTHER OUTCOMES:
Comparison of Fungal-Free | Day 14 (±1 day), Day 28 (±1 day), Day 60 (±5 days), and Day 120 (±7 days)
  The number of subjects in each treatment group who are fungal-free.
Comparison of Fungal-Free | Day 14 (±1 day), Day 28 (±1 day), Day 60 (±5 days), and Day 120 (±7 days)
  The percentage of subjects in each treatment group who are fungal-free.
Comparison of Presence and Severity of GHVD | Day 90 (±7 days)
  Evaluate the presence and severity of GVHD in subjects randomized to Rezafungin for Injection compared to the SAR.
Comparison of Fungal-Free with AML | Day 90 (±7 days)
  The number of subjects in each treatment group who are fungal-free with an underlying diagnosis of acute myeloid leukemia (AML).
Comparison of Fungal-Free with AML | Day 90 (±7 days)
  The percentage of subjects in each treatment group who are fungal-free with an underlying diagnosis of acute myeloid leukemia (AML).
Compare Incidence of IFD | Day 14 (±1 day), Day 28 (±1 day), Day 60 (±5 days), Day 90 (±7 days), and Day 120 (±7 days)
  Evaluate the incidence of proven, probable, possible, and presumptive IFD in subjects randomized to Rezafungin for Injection compared to the SAR.
Compare Relapse-Free Survival | Day 1 through follow-up visit (Day 120)
  Evaluate relapse-free survival, with and without adjustment for patient comorbidity indices, in subjects randomized to Rezafungin for Injection compared to the SAR.
Evaluate PK (Cmax) | Day 0 (±2 days) within 10 minutes before end of infusion, and one sample between end of infusion and 12 hours after end of infusion; Days 1-4, one sample at any time; Day 7 (±1 day), Day 28 (±1 day), and Day 63 (±1 day) prior to dosing; and EOT visit
  Evaluate maximum plasma concentration (Cmax).
Evaluate PK (Tmax) | Day 0 (±2 days) within 10 minutes before end of infusion, and one sample between end of infusion and 12 hours after end of infusion; Days 1-4, one sample at any time; Day 7 (±1 day), Day 28 (±1 day), and Day 63 (±1 day) prior to dosing; and EOT visit
  Evaluate time to Cmax.
Evaluate PK (AUC) | Day 0 (±2 days) within 10 minutes before end of infusion, and one sample between end of infusion and 12 hours after end of infusion; Days 1-4, one sample at any time; Day 7 (±1 day), Day 28 (±1 day), and Day 63 (±1 day) prior to dosing; and EOT visit
  Evaluate area under the curve (AUC).
Compare Post-Engraftment Cytopenias and Transfusion Requirements | Day 1 through follow-up visit (Day 120)
  Evaluate post-engraftment cytopenias and transfusion requirements of Rezafungin for Injection compared to the SAR.
Compare Infections Caused by TMP/SMX-Sensitive Organisms | Day 14 (±1 day), Day 28 (±1 day), Day 60 (±5 days), Day 90 (±7 days), and Day 120 (±7 days)
  Evaluate infections caused by TMP/SMX-sensitive organisms (Toxoplasma gondii [T. gondii], Nocardia spp.) in Rezafungin for Injection compared to the SAR.
Compare Antifungal Prophylaxis | Day 14 (±1 day), Day 28 (±1 day), Day 60 (±5 days), Day 90 (±7 days), and Day 120 (±7 days)
  Evaluate interruption and discontinuation of antifungal prophylaxis due to suspected IFDs of Rezafungin for Injection compared to the SAR.
Compare the health economics outcome research (HEOR) variable of "Days in Hospital" | Once weekly for outpatient, or twice weekly for inpatient, at completion of study drug therapy [Day 90 (±7 days)] and for 30 days [Day 120 (±7 days)]
  Evaluate the number of hospital days for subjects randomized to Rezafungin for Injection compared to the SAR.
Compare the health economics outcome research (HEOR) variable of "Days in Intensive Care Unit (ICU)" | Once weekly for outpatient, or twice weekly for inpatient, at completion of study drug therapy [Day 90 (±7 days)] and for 30 days [Day 120 (±7 days)]
  Evaluate the number of days in ICU for subjects randomized to Rezafungin for Injection compared to the SAR.
Compare the health economics outcome research (HEOR) variable of "Readmission due to Infectious Disease Diagnosis" | Once weekly for outpatient, or twice weekly for inpatient, at completion of study drug therapy [Day 90 (±7 days)] and for 30 days [Day 120 (±7 days)]
  Evaluate readmission(s) due to infectious disease diagnosis for subjects randomized to Rezafungin for Injection compared to the SAR.
Compare the health economics outcome research (HEOR) variable of "Readmission due to Invasive Fungal Disease Diagnosis" | Once weekly for outpatient, or twice weekly for inpatient, at completion of study drug therapy [Day 90 (±7 days)] and for 30 days [Day 120 (±7 days)]
  Evaluate readmission(s) due to invasive fungal disease diagnosis for subjects randomized to Rezafungin for Injection compared to the SAR.
Compare the health economics outcome research (HEOR) variable of "Alternative Antifungal Therapy" | Once weekly for outpatient, or twice weekly for inpatient, at completion of study drug therapy [Day 90 (±7 days)] and for 30 days [Day 120 (±7 days)]
  Evaluate the incidence of alternative antifungal therapy compared to Rezafungin for Injection and the SAR.
Compare the health economics outcome research (HEOR) variable of "Antibiotic Therapy" | Once weekly for outpatient, or twice weekly for inpatient, at completion of study drug therapy [Day 90 (±7 days)] and for 30 days [Day 120 (±7 days)]
  Evaluate the incidence of antibiotic therapy compared to Rezafungin for Injection and the SAR.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Cox, PhD, Study Director — Mundipharma Research Limited
Locations (53):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCLA Center for Health Sciences, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Augusta University Medical Center, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - John Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Physicians, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mary Hitchcock Memorial Hospital Dartmouth-Hitchcock, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Stony Brook University Hospital, Stony Brook, New York
  - The University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - VCU Medical Center Main Hospital, Richmond, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Belgium (2):
  - AZ Sint-Jan, Bruges, West Vlaanderen
  - University Hospitals Leuven, Campus Gasthuisberg - UZ Leuven, Leuven
- Canada (2):
  - Hamilton Health Sciences' Juravinski Hospital, Hamilton
  - McGill University Health Center, Montreal
- France (8):
  - Jean Minjoz Hospital, Besançon
  - Henri Mondor Hospital, Créteil
  - Grenoble Alpes University Hospital Center, Grenoble
  - University Hospital of Limoges, Limoges
  - University Hospital of Nantes, Nantes
  - Hospital Saint Antoine Ap-Hp, Paris
  - University Hospital of Bordeaux, Pessac
  - Lyon-Sud Hospital Center, Pierre-Bénite
- Germany (5):
  - University Hospital of Cologne, Cologne
  - University Hospital Carl Gustav Carus Dresden, Dresden
  - Johannes Gutenberg University Medical Center, Mainz
  - University Hospital Münster, Münster
  - University Hospital Wurzburg UKW, Würzburg
- Italy (4):
  - San Martino Polyclinic Hospital, Genova
  - IEO Istituto Europeo di Oncologia, Milan
  - Agostino Gemelli University Policlinic, Rome
  - Humanitas Cancer Center, Rozzano
- Spain (8):
  - University Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic of Barcelona, Barcelona
  - University Hospital Ramon y Cajal, Madrid
  - Puerta de Hierro Majadahonda University Hospital, Majadahonda
  - University Hospital of Salamanca, Salamanca
  - University Hospital Marques de Valdecilla, Santander
  - University Hospital of Valencia, Valencia
  - La Fe University and Polytechnic Hospital, Valencia
- University Hospitals Geneva, Geneva, Switzerland
- United Kingdom (5):
  - Addenbrookes Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Kings College Hospital NHS Foundation Trust, London
  - St. George's University Hospitals NHS Foundation Trust, London
  - The Royal Marsden Nhs Foundation Trust, London

REFERENCES:
- [Derived] Cross SJ, Wolf J, Patel PA. Prevention, Diagnosis and Management of Pneumocystis jirovecii Infection in Children With Cancer or Receiving Hematopoietic Cell Therapy. Pediatr Infect Dis J. 2023 Dec 1;42(12):e479-e482. doi: 10.1097/INF.0000000000004102. Epub 2023 Sep 21. No abstract available. PMID 37773627
- [Derived] Ham YY, Lewis JS 2nd, Thompson GR 3rd. Rezafungin: a novel antifungal for the treatment of invasive candidiasis. Future Microbiol. 2021 Jan;16(1):27-36. doi: 10.2217/fmb-2020-0217. PMID 33438477